CLINICAL TRIAL: NCT05922475
Title: Neither Pre-sleep Nor Post-exercise Protein Consumption Influences Resistance Exercise Training Adaptations in Older Adults
Brief Title: Efficacy of Pre-sleep or Post-exercise Protein During 12 Weeks of Resistance Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Alexander Klemp, Principal investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25996
Record Dates: First submitted 2023-05-27; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Aging
Keywords: Exercise; Hypertrophy; Strength; Power
MeSH Terms: conditions — Motor Activity; Hypertrophy | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post-exercise protein (Experimental): Consumed 40 g of supplemental protein immediately after exercise sessions and in between breakfast and lunch on non-exercise days.
  Interventions: Dietary Supplement: Protein
- Pre-sleep protein (Experimental): Consumed 40 g of supplemental protein 30 minutes before sleep every day.
  Interventions: Dietary Supplement: Protein
- Resistance exercise training only (Placebo Comparator): Did not consume supplemental protein.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Protein — Post-exercise protein group consumed protein immediately after exercise sessions.
  Pre-sleep protein group consumed protein 30 minutes before sleep.
  Arms: Post-exercise protein; Pre-sleep protein
Other: Placebo — Resistance exercise training only group did not consume supplemental protein.
  Arms: Resistance exercise training only

SUMMARY:
The goal of this clinical trial is to compare the effects of protein consumption before sleep or immediately after exercise during 12 weeks of resistance exercise training in older adults. The main questions it aims to answer are:

Are there differences in muscle growth or strength during 12 weeks of resistance training when 40 grams of protein is consumed either before sleep or immediately after exercise? Are there differences in cognitive performance during 12 weeks of resistance training when 40 grams of protein is consumed either before sleep or immediately after exercise?

This study is a randomized double-blind placebo-controlled study. Participants will be randomly allocated into 1 of 3 groups. All three groups will perform the same 12-week resistance exercise training program two times per week and consume 40 g of protein: 1) Immediately post-exercise, 2) 30 minutes prior to sleep, or 3) no supplemental protein (control). Test of muscle growth and strength, and cognitive performance will be measure before, during, and after the exercise training program.

Researchers will compare the 3 conditions to determine if consume protein after exercise or before sleep during 12 weeks of resistance exercise training affects muscle growth and strength, and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Male between 60-75 years old at the time of enrollment.

Exclusion Criteria:

* Diagnosis of cardiac or peripheral vascular disease
* Stroke, kidney dysfunction
* Metabolic disease
* Uncontrolled hypertension
* Orthopedic limitations
* Skeletal muscle complications
* Milk allergy
* Psychiatric conditions
* Use of psychotropic drugs
* Cognitive impairment (scoring 26 points or less on the Montreal Cognitive Assessment)
* Participation in a structured regular exercise program within the past 6 months
* Actively attempting to increase or decrease body mass
* Body mass index (BMI) of ≥ 35 kg/m2

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | Week 0, 6, and 12
  Change in muscle thickness of the quadriceps muscles in centimeters from week 0 (baseline) to week 6 (midpoint) to week 12 (end of study).

SECONDARY OUTCOMES:
Maximum muscular strength | Week 0, 6, and 12
  Changes in strength of the chest press and leg press exercises in kilograms from week 0 (baseline) to week 6 (midpoint) to week 12 (end of study).
Muscle power | Week 0, 6, and 12
  Changes in power (Watts) during a sit-to-stand task from week 0 (baseline) to week 6 (midpoint) to week 12 (end of study).
Cognitive performance | Week 0 and 12
  Changes in the number of correct responses during the digit symbol substitution task and pattern comparison tests from week 0 (baseline) to week 12 (end of study).
Measures associated appetite | Week 0, 6, and 12
  Changes in subjective measures of hunger, satiety, and desire to eat on a 0-100 millimeter (higher values indicating stronger feeling) visual analog scale from week 0 (baseline) to week 6 (midpoint) to week 12 (end of study).
Total sleep time | Week 0 and 12
  Changes in actigraphy watch measured total sleep time in hours from week 0 (baseline) to week 12 (end of study).
Sleep latency | Week 0 and 12
  Changes in actigraphy watch measured sleep latency in minutes from week 0 (baseline) to week 12 (end of study).
Measures associated with sleep | Week 0 and 12
  Changes in actigraphy watch measured sleep efficiency (ratio of time spent asleep to the time spent in bed) in percentage from week 0 (baseline) to week 12 (end of study).
Nitrogen balance | Week 0 and 12
  Changes in urinary nitrogen balance (grams per day) from week 0 (baseline) to week 12 (end of study).
Free insulin-like growth factor 1 | Week 0 and 12
  Changes in plasma free insulin-like growth factor 1 concentration (nanogram per deciliter) from week 0 (baseline) to week 12 (end of study).
Mood | Week 0 and 12
  Changes in the Profile of Mood State rating scale categories of tension, depression, anger, fatigue, confusion, vigor, and total mood disturbance from week 0 (baseline) to week 12 (end of study) via a 1 to 5 scale (higher score indicates stronger feeling).

CONTACTS AND LOCATIONS:
Overall Officials: Alex O Klemp, PhD, Principal Investigator — Student
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klemp AO, Ormsbee MJ, Yeh M, Sokolowski CM, Kim DH, Panton LB, Kim JS. Neither pre-sleep nor post-exercise protein consumption influences resistance exercise training adaptations in older adults. J Int Soc Sports Nutr. 2025 Dec;22(1):2519511. doi: 10.1080/15502783.2025.2519511. Epub 2025 Jun 20. PMID 40539259

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05922475/Prot_SAP_ICF_000.pdf